CLINICAL TRIAL: NCT03149185
Title: Technology Based Psychosocial Intervention for Symptom Management and HRQOL in Men Living With Advanced Prostate Cancer
Acronym: PC-CHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00064136
Record Dates: First submitted 2017-04-19; First posted 2017-05-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; advanced prostate cancer; technology based
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized experimental trial designed to evaluate the effects of a 10-week technology-based group cognitive-behavioral stress management intervention (T-CBSM) vs. a health promotion (T-HP) group-based attention matched control condition. This is a 2 x 3 design with group assignment (T-CBSM vs. T-HP) as the between group factor, and time (baseline [T1], 6-months post-T1 [T2], and 12-months post T1 [T3]) as the within-group factor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-CBSM (Active Comparator): Technology based cognitive behavioral stress management.
  Interventions: Behavioral: Technology based cognitive behavioral stress management
- T-HP (Active Comparator): Technology based health promotion (control condition)
  Interventions: Behavioral: Technology based health promotion group-based attention matched control condition

INTERVENTIONS:
Behavioral: Technology based cognitive behavioral stress management — Intervention is delivered through Telecare (web based technology) in a group for 60-90 minutes/session. During each session, participants are taught/discuss a new anxiety/arousal reduction technique and focus on stress management. Efficacy of available treatments, disease course, symptom burden, communication with intimate partner and/or family members and health care provider, impact of stress on physical and mental health and symptoms, and management of APC and HT symptoms are used for educational purposes and as catalysts for discussing TCBSM techniques. We allow participants to describe psychosocial stressors with an emphasis on symptoms and disruption, HRQOL and their coping responses for in-session role-plays. Participants are able to access the system at any time to retrieve relaxation and stress management didactics, and contact community resources and other participants in their group.
  Other Names: T-CBSM
  Arms: T-CBSM
Behavioral: Technology based health promotion group-based attention matched control condition — Sessions include content from relevant NCI, ACS and other resources developed to address the needs of advanced cancer populations into each topic session. All sessions address APC-specific issues. While men receiving treatment for APC remain interested in general health issues and as they become increasingly aware of the end-of-life issues raised by facing advanced disease, they seem to be interested in making life changes in areas in which they do exercise control (e.g., nutrition), and as such have been integrated into the T-HP modules in addition to general recommendations from sources such as American Heart Association, the NIA and the ACS. T-HP participants are scheduled for weekly group-based health information and promotion sessions (60-90 mins.), which are delivered via our videophones by our T-HP facilitators.
  Other Names: T-HP
  Arms: T-HP

SUMMARY:
The purpose of this study is to examine the effects of various factors such as emotions, stress, stress management techniques (for example relaxation and coping techniques), and health information on quality of life, distress, depression, coping, and physical health in men diagnosed with advanced prostate cancer. The investigators also evaluate the effectiveness of a 10-week group-based internet delivered psychosocial intervention. Primary outcomes are symptom burden (e.g., urinary function, fatigue, pain) and HRQOL (e.g., general, physical & social functioning).

Participation in this study includes three face-to-face assessments: baseline (at the beginning of the research study), 6-month follow-up, and 12-month follow-up. The 6- and 12-month follow-up interviews are conducted after the participant has completed the 10-week group intervention. Participants are randomized into either an intervention group (targets stress management skills - relaxation, coping) or a control group (health information and health promotion strategies - benefits of proper nutrition and treatment compliance). Both groups meet for 10 consecutive weeks through an internet video conferencing platform.

At the baseline, 6- and 12-month follow-ups, the investigators collect blood and saliva samples. The blood samples go through a three-day process in which the investigators extract and store serum, plasma, and cells for further analysis and gather proliferation data. The investigators use the saliva to measure the cortisol diurnal rhythm.

DETAILED DESCRIPTION:
This 5-year study evaluates the effects of a 10-week technology-based and delivered cognitive-behavioral stress management intervention (T-CBSM) on symptom burden in men with advanced prostate cancer (APC) undergoing hormonal therapy (HT), or HT with prior radiotherapy (RT) and/or radical prostatectomy (RP). APC is chronic and debilitating with survival rates about 32% and even lower rates for ethnic minorities. Most (70%) men diagnosed with APC receive HT to control progression. HT is associated with side effects including depression, fatigue, hot flashes, and sexual and urinary dysfunction, while RT and RP also lead to fatigue, irritation, urinary dysfunction, etc. Symptoms combined with challenges of living with advanced disease (e.g., unpredictable disease course) significantly deteriorate health-related quality of life (HRQOL). Yet, there is limited information on how psychosocial factors impact symptom burden, or on the efficacy of psychosocial interventions in reducing symptom burden and improving HRQOL. Furthermore, psychosocial modulation of endocrine and immune function is associated with symptoms and HRQOL in cancer patients, including those with advanced disease. Stress-related disruption in diurnal cortisol can promote inflammation that can exacerbate symptoms (e.g., fatigue, depression, pain). In the investigaros' pilot work, the investigators observed that audio-based T-CBSM improves social and physical functioning, and decreases symptom burden in APC. Moreover, targets of T-CBSM (e.g., coping skills) explain reductions in symptoms, whereas decreases in inflammatory cytokines (e.g., IL-1, IL-6) and enhanced cortisol regulation are associated with decreases in symptoms such as depression, pain, urinary dysfunction and fatigue. The investigators propose to deliver an enhanced T-CBSM intervention to (a) capitalize on new technology using a video-conferencing for hard-to-reach and ethnically diverse patients, (b) incorporate a neuroimmune model of symptom regulation and management, and (c) test the efficacy of Web-CBSM in a multi-ethnic sample of 200 men living with APC. Men will be randomized to a T-CBSM group intervention or a health promotion group (T-HP) control condition. The investigators' primary aims are to determine the extent to which randomization to T-CBSM relative to T-HP is associated with: (Aim 1) improved symptom burden management and HRQOL, (Aim 2) reduced distress and interpersonal disruption, and improved stress management skills, and (Aim 3) improved neuroimmune regulation (i.e., normalized diurnal cortisol & decreases in inflammatory cytokines). The investigators will also test (Aim 4) a set of hypothesized pathways (e.g., T-CBSM driven changes in distress, stress management skills, neuroimmune regulation, etc.) that explain the association between group assignment and the primary outcomes of symptom burden and HRQOL. This is a 2x3 randomized experimental design with condition (T-CBSM vs. T-HP) as the between groups factor and time (baseline [T1], 6-mos. post-baseline [T2], & 12-mos. post-baseline [T3]) as the within groups factor.

Experimental Design. This is a randomized experimental trial designed to evaluate the effects of a 10-week technology-based group cognitive-behavioral stress management intervention vs. a health promotion group-based attention matched control condition. Primary outcomes are symptom burden (e.g., urinary function, fatigue, pain) and HRQOL (e.g., general, physical & social functioning).

Participants. Participants will be 200 ethnically diverse men ages 50 or older, with stage III or IV prostate cancer (i.e., APC) who are on hormonal treatment (HT; androgen ablation, androgen deprivation, chemical castration) with or without radiotherapy (RT). Participants must also have undergone HT within the past 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years of age
* Fluent in spoken English (6th grade level required to complete assessments and participate in groups)
* Diagnosis of Stage III or IV (T3/N1/ M0-T4/N3/M1) prostate cancer
* Received HT, or HT and RT treatment within the past year or is currently receiving HT, or HT and RT
* Some patients with prior inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis) may be enrolled, per P.I. discretion, based on a case-by-case review
* Willingness to be randomized and followed for 12 months

Exclusion Criteria:

* Received treatment for a type of cancer other than prostate or skin cancer within the past 5 years or is currently receiving treatment for a cancer other than prostate or skin
* Prior inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis), as these conditions can interfere with adequate participation in our experimental conditions may be exclusionary, per P.I. discretion, based on a case-by-case review
* Active alcohol abuse or dependence OR inpatient treatment for alcohol abuse within the last 6 months may be exclusionary, per P.I. discretion
* Active substance abuse or dependence OR inpatient treatment for substance abuse within the last 6 months may be exclusionary, per P.I. discretion
* Acute or chronic immune system medical conditions, medications or other conditions that impact immune and endocrine function (e.g., CFS, Lupus, rheumatoid arthritis, Sjogren's disease, SLE, Hepatitis C, or any immunosuppressive treatment requiring conditions)
* Life expectancy <12 months.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
Change in symptom burden from baseline (T1) to 6- and 12-month follow-up assessments (T2 & T3) relative to participants in T-HP (control). | baseline (T1), 6-months post-baseline (T2), and 12-months post-baseline (T3)
  Symptom burden will be measured with the Expanded PC Index Composite (EPIC)
Change in HRQOL from baseline (T1) to 6- and 12-month follow-up assessments (T2 & T3) relative to participants in T-HP (control). | baseline (T1), 6-months post-baseline (T2), and 12-months post-baseline (T3)
  SF-12, a short form version of the commonly used SF-36, a health survey designed to assess multiple dimensions of HRQOL

OTHER OUTCOMES:
Distress & Positive/Negative Affect | baseline (T1), 6-months post-baseline (T2), and 12-months post-baseline (T3)
  Memorial Anxiety Scale for Prostate Cancer patients (MAX-PC), an 18-item instrument that detects symptoms of anxiety in PC patients.
Interpersonal Disruption | baseline (T1), 6-months post-baseline (T2), and 12-months post-baseline (T3)
  The sum of two scales from the Sickness Impact Profile (SIP)cviii, Recreation and Pastimes and Social interactions.
Stress Management Skills | baseline (T1), 6-months post-baseline (T2), and 12-months post-baseline (T3)
  Stress awareness, cognitive appraisals, relaxation skills, coping and communication skills, and interpersonal skills will be assessed using the Measure of Current States (MOCS)
Neuroimmune Regulation | baseline (T1), 6-months post-baseline (T2), and 12-months post-baseline (T3)
  Salivary Cortisol & Inflammatory Cytokines

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benzo RM, Moreno PI, Fox RS, Silvera CA, Walsh EA, Yanez B, Balise RR, Oswald LB, Penedo FJ. Comorbidity burden and health-related quality of life in men with advanced prostate cancer. Support Care Cancer. 2023 Jul 28;31(8):496. doi: 10.1007/s00520-023-07962-6. PMID 37501020
- [Derived] Walsh EA, Boland CL, Popok PJ, Pedreira PB, Fox RS, Moreno PI, Yanez B, Penedo FJ. Marital status and perceived stress in men with advanced prostate cancer: A randomized-controlled trial of cognitive behavioral stress management. J Psychosom Res. 2023 Apr;167:111198. doi: 10.1016/j.jpsychores.2023.111198. Epub 2023 Feb 16. PMID 36812663
- [Derived] Walsh EA, Pedreira PB, Moreno PI, Popok PJ, Fox RS, Yanez B, Antoni MH, Penedo FJ. Pain, cancer-related distress, and physical and functional well-being among men with advanced prostate cancer. Support Care Cancer. 2022 Dec 14;31(1):28. doi: 10.1007/s00520-022-07453-0. PMID 36515785
- [Derived] Penedo FJ, Fox RS, Oswald LB, Moreno PI, Boland CL, Estabrook R, McGinty HL, Mohr DC, Begale MJ, Dahn JR, Flury SC, Perry KT, Kundu SD, Yanez B. Technology-Based Psychosocial Intervention to Improve Quality of Life and Reduce Symptom Burden in Men with Advanced Prostate Cancer: Results from a Randomized Controlled Trial. Int J Behav Med. 2020 Oct;27(5):490-505. doi: 10.1007/s12529-019-09839-7. PMID 31898309
- [Derived] Fox RS, Moreno PI, Yanez B, Estabrook R, Thomas J, Bouchard LC, McGinty HL, Mohr DC, Begale MJ, Flury SC, Perry KT, Kundu SD, Penedo FJ. Integrating PROMIS(R) computerized adaptive tests into a web-based intervention for prostate cancer. Health Psychol. 2019 May;38(5):403-409. doi: 10.1037/hea0000672. PMID 31045423